CLINICAL TRIAL: NCT06912503
Title: Comparative Analysis About the Dimensional Accuracy of Diagnostic Trial Restoration Transferring Performed With Four Different Methods for Trial Restoration Matrix Fabrication: an in Vivo Study
Brief Title: Comparison of Trial Restoration Matrix Fabrication Methods
Status: Completed | Type: Observational
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Sponsor
Other Study IDs: REST-ECL-2020-03
Record Dates: First submitted 2025-03-21; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-01

CONDITIONS: Teeth Restoration
Keywords: Restoration of worn teeth

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Condensation silicone matrix: base and catalyst paste, 85 Shore A (Zetalabor, Zhermack) were mixed and applied over the waxing printed cast ensuring an overall even distribution of the material buccally and incisally over the cast guaranteeing a minimal thickness of 8-10mm. The setting time advised by the fabricant was respected. After, the condensation silicone matrix was measured, marked and trimmed, using a dental model trimmer (Dual wheel dental model trimmer, Dentaurum Inc.) to obtain a 6 mm thickness of the matrix. Finally, a vacuum shell was fabricated over the final volume of the condensation silicone matrix to replicate the material distribution and thickness for the fabrication of the other matrixes.
  Interventions: Device: Device to deliver trial restoration matrix
- Addition PVS-silicone matrix: a two-step putty wash addition silicone technique was adopted using poly-vinylsiloxane material, 60 Shore A (Aquasil, Dentsply Sirona). First a spacer was applied over the printed waxed cast and the putty silicone was packed inside the previously fabricated vacuum shell. After the setting time advised by the fabricant, the matrix and the spacer were removed from the cast and the light silicone was poured to reline the waxed cast. Once set the PVS-silicone matrix was removed from the vacuum shell and the interproximal areas trimmed using a scalpel. Finally, a layer of resin-based shell (Triad light-curing trays, Dentsply) was applied and cured over the PVS silicone matrix.
  Interventions: Device: Device to deliver trial restoration matrix
- Transparent addition PVS-silicone matrix: the PVS-silicone, 53 Shore A (Elite glass, Zhermack) poured inside the vacuum shell previously fabricated and relined over the waxed cast. After the setting time advised by the fabricant the cast was removed and a hole was performed incisally to each waxed tooth using a bur in order to insert a tip of flowable composite resin.
  Interventions: Device: Device to deliver trial restoration matrix
- CAD/CAM combination matrix: First, a 3D printed resin matrix was designed (Exocad DentalCAD; Exocad GmbH) and printed (Phrozen Mini 4K, Phrozen Technology) using a clear biocompatible resin (Dental Clear, Harz Labs) providing a calibrated and equally distributed space for the PVS-silicone material, which reproduced the diagnostic waxed design. Later a low-shore PVS-silicone material, 60 Shore A (Aquasil light, Dentsply Sirona) was used to reline the AM matrix. The rigid matrix would guide the relining process thanks to dental-supported distal stops and buccal openings for visual assessment of proper fitting.
  Interventions: Device: Device to deliver trial restoration matrix

INTERVENTIONS:
Device: Device to deliver trial restoration matrix — Auto-polymerization bisacrylic material (Luxatemp Star, DMG) was used to perform the trial restoration for condensation silicone matrix, addition PVS-silicone matrix with external resin-based shell and CAD/CAM combination matrix. Light-cured flowable composite-resin (Filtek Flow, 3M Dental Products) was used to perform the trial restoration for transparent addition PVS-silicone matrix. The rationale behind using different material stands on the material selection usually chosen by clinicians for each matrix.
  In the same appointment 4 trial restorations were performed to each patient using the four different matrixes.

SUMMARY:
This observational analytical in vivo study aimed to assess the dimensional accuracy of diagnostic trial restorations fabricated through four different techniques: condensation silicone matrix without external shell, addition polyvinylsiloxane (PVS)-silicone matrix with an external resin-based shell, transparent addition PVS-silicone matrix with an external vacuum shell, and a CAD/CAM combination matrix.

Methods: Patients (n=20) in need of anterior upper teeth aesthetic rehabilitation were recruited. Clinical and radiographic examinations, intraoral scanning, and dental CAD software were used to design a virtual diagnostic waxing. A 3D printed waxed cast was obtained, and four different matrices were fabricated. Trial restorations were performed using calibrated materials, and intraoral scans were taken for each restoration. Linear and volumetric discrepancies were evaluated using reverse engineering alignment software

DETAILED DESCRIPTION:
The present study was an observational analytical in vivo study approved by the CEIM (Comité de Ética de Investigación con Medicamentos) of the International University of Catalunya.

The patient recruitment was carried out among patients from the Clínica Universitaria Odontológica (CUO) in need of an aesthetic rehabilitation of the anterior upper teeth.

The inclusion and exclusion criteria of the sample were the following:

Inclusion Criteria

* Patients between 18 and 70 years old.
* Patients who maintain the six upper anterior teeth.
* Patients in need of an additive restorative rehabilitation. Exclusion Criteria
* Patients with removable prostheses.
* Patients with an absent upper anterior tooth.
* Patients with a buccal inclination of any of the six upper anterior teeth.

All the information of the study was delivered to the patients before signing and obtaining the inform consent form.

Study design Each patient underwent a primary diagnostic phase, which included clinical and radiographic examinations, extraoral and intraoral photography and intraoral scanning (IOS) (Trios3, 3Shape) to obtain standard tessellation language (STL) files. STL files were imported into a dental CAD (computed assisted design) software (Exocad DentalCAD; Exocad GmbH) to design a virtual diagnostic waxing for the 6 maxillary anterior teeth. The CAD design was performed by the same operator for each case and a resin-printed cast of the waxing was fabricated using additive manufacturing (AM) technology with a 3D printing machine (Phrozen Mini 4K, Phrozen Technology) using model resin (Aqua-Gray 4K printer resin, Phrozen Technology). The 3D printed waxed cast was introduced into an ultrasonic alcohol bath (96%) for 5 minutes, dried and cured in an ultraviolet curing chamber (7 minutes and 7 minutes submerged in glycerine gel) (Wash & Cure machine 2.0, Anycubic 3D Printing).

Each diagnostic waxed printed cast was then digitized using the same intraoral scanning (Trios3, 3Shape) to obtain the reference model STL files used as control group for the study.

Four different types of matrixes were fabricated from the diagnostic waxing printed cast by the same operator: condensation silicone matrix, addition PVS-silicone matrix with external resin-based shell, transparent addition PVS-silicone matrix with external vacuum shell, and a CAD/CAM (computer assisted machining) combination matrix.

Condensation silicone matrix: base and catalyst paste, 85 Shore A (Zetalabor, Zhermack) were mixed and applied over the waxing printed cast ensuring an overall even distribution of the material buccally and incisally over the cast guaranteeing a minimal thickness of 8-10mm. The setting time advised by the fabricant was respected. After, the condensation silicone matrix was measured, marked and trimmed, using a dental model trimmer (Dual wheel dental model trimmer, Dentaurum Inc.) to obtain a 6 mm thickness of the matrix.

Finally, a vacuum shell was fabricated over the final volume of the condensation silicone matrix to replicate the material distribution and thickness for the fabrication of the other matrixes.

Addition PVS-silicone matrix: a two-step putty wash addition silicone technique was adopted using poly-vinylsiloxane material, 60 Shore A (Aquasil, Dentsply Sirona). First a spacer was applied over the printed waxed cast and the putty silicone was packed inside the previously fabricated vacuum shell. After the setting time advised by the fabricant, the matrix and the spacer were removed from the cast and the light silicone was poured to reline the waxed cast. Once set the PVS-silicone matrix was removed from the vacuum shell and the interproximal areas trimmed using a scalpel. Finally, a layer of resin-based shell (Triad light-curing trays, Dentsply) was applied and cured over the PVS silicone matrix.

Transparent addition PVS-silicone matrix: the PVS-silicone, 53 Shore A (Elite glass, Zhermack) poured inside the vacuum shell previously fabricated and relined over the waxed cast. After the setting time advised by the fabricant the cast was removed and a hole was performed incisally to each waxed tooth using a bur in order to insert a tip of flowable composite resin.

CAD/CAM combination matrix: First, a 3D printed resin matrix was designed (Exocad DentalCAD; Exocad GmbH) and printed (Phrozen Mini 4K, Phrozen Technology) using a clear biocompatible resin (Dental Clear, Harz Labs) providing a calibrated and equally distributed space for the PVS-silicone material, which reproduced the diagnostic waxed design. Later a low-shore PVS-silicone material, 60 Shore A (Aquasil light, Dentsply Sirona) was used to reline the AM matrix. The rigid matrix would guide the relining process thanks to dental-supported distal stops and buccal openings for visual assessment of proper fitting.

Auto-polymerization bisacrylic material (Luxatemp Star, DMG) was used to perform the trial restoration for condensation silicone matrix, addition PVS-silicone matrix with external resin-based shell and CAD/CAM combination matrix. Light-cured flowable composite-resin (Filtek Flow, 3M Dental Products) was used to perform the trial restoration for transparent addition PVS-silicone matrix. The rationale behind using different material stands on the material selection usually chosen by clinicians for each matrix.

In the same appointment 4 trial restorations were performed to each patient using the four different matrixes. The intraoral scan STL file, previously recorded in the diagnostic appointment, was duplicated and the area corresponding to the 6 anterior teeth was trimmed virtually, this procedure was executed 4 times. Each trial restoration was performed and then scanned over the trimmed STL files.

A total of 100 STL files were acquired. Four intraoral scans per group were obtained for each patient. The control group was the intraoral scan of the printed waxed cast which was used as a reference STL file.

The accuracy of each technique was calculated from the discrepancy between the IOS of each trial restoration scan and the reference STL.

Each trial restoration IOS (addition, condensation, clear, combined) was imported and aligned to the control reference STL cast of the waxed printed cast using the "best fit" algorithm of a non-dental reverse engineering software (Cx Geomagic Control X). Volumetric discrepancies, limited to the diagnostic waxing area, were measured using the RMS value. Linear discrepancies were calculated measuring the distance in 4 points (cervical, medial, lower medial and incisal) on the buccal aspect of each waxed tooth, from 13 to 23, between the trial restoration STL file and the control STL file.

All the measurements were recorded into an Excel page.

Statistical analysis After analyzing normality, Levene's test will be used to demonstrate wether there is a statistically significant difference amongst the measured linear and volumetric discrepancies' standard deviations (p<0.05) or not. Non-parametric Kruskal-Wallis (K-W) and Mann-Whitney (M-W) tests will be performed to assess statistical differences in the linear and volumetric discrepancies in the studied groups Statistical significance will be set at p<0.05 with a confidence interval of 95%.

ELIGIBILITY:
* Patients between 18 and 70 years old.
* Patients who maintain the six upper anterior teeth.
* Patients in need of additive restorative rehabilitation. Exclusion Criteria
* Patients with removable prostheses.
* Patients with an absent upper anterior tooth.
* Patients with a buccal inclination of any of the six upper anterior teeth.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients attending the university dental clinic
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-01-08 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
Volumetric discrepancy | From enrollment the patient underwent the different procedures within a month. The four procedures were delivered to the patient the same day, one after the other, in an order determined by the randomization
  . Each trial restoration IOS (addition, condensation, clear, combined) was imported and aligned to the control reference STL cast of the waxed printed cast using the "best fit" algorithm of a non-dental reverse engineering software (Cx Geomagic Control X). Volumetric discrepancies, limited to the diagnostic waxing area, were measured using the RMS value.

CONTACTS AND LOCATIONS:
Overall Officials: MIGUEL ROIG CAYON, MD, DDS, Study Chair — Universitat Internacional de Catalunya
Locations (1):
- Universitat Internacional de Catalunya, Barcelona, BARCELONA, Spain

IPD SHARING:
Plan to Share IPD: Yes
All documentation of the study will be included in a publication planned to be published at the end of the study. After that, all the information (study protocol, informed consent, results) will be uploaded in a public repository from UIC
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Start date: September 2025
Access Criteria: Open access